CLINICAL TRIAL: NCT01572987
Title: Endoscopic Resection or Ablation for Patients With Dysplasia or Intramucosal Cancer in Barrett's Esophagus
Brief Title: Endoscopic Resection or Ablation for Patients With Dysplasia or Cancer Requiring Treatment of Barrett's Esophagus
Acronym: ERADICATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment goals not being met
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); Cook Group Incorporated (Industry); Washington University School of Medicine (Other); Columbia University (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS0058
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Barrett's Esophagus; Esophageal Neoplasms
Keywords: Barrett's Esophagus; Esophageal neoplasms; Radiofrequency ablation; Endoscopic mucosal resection
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA arm (Active Comparator): Under this arm, study patients will undergo radiofrequency ablation.
  Interventions: Device: Radiofrequency Ablation(RFA) by HALO device.
- EMR arm (Active Comparator): Under this arm, the individuals will undergo endoscopic mucosal resection.
  Interventions: Device: Endoscopic mucosal resection(EMR) by mucosectomy kit.

INTERVENTIONS:
Device: Radiofrequency Ablation(RFA) by HALO device. — RFA or Surveillance every 2 months for 1 year.
  Other Names: HALO Ablation Technology(BÂRRX Medical, Inc).
  Arms: RFA arm
Device: Endoscopic mucosal resection(EMR) by mucosectomy kit. — EMR or surveillance every 2 months.
  Other Names: Duette multi-band mucosectomy kit (Cook Medical).
  Arms: EMR arm

SUMMARY:
This clinical trial will evaluate a patient population with Barrett's esophagus(BE) containing high grade dysplasia or intramucosal cancer and compare the effects of endoscopically-guided radiofrequency ablation system(RFA) and endoscopically-guided stepwise endoscopic mucosal resection(S-EMR).

DETAILED DESCRIPTION:
This is a multi-center prospective, randomized controlled trial conducted at 4 centers. The patients with high grade dysplasia(HGD) and/or esophageal cancer(EC) who meet the study criteria will be enrolled, undergo a baseline diagnostic EMR and then be randomized in a 1:1 ratio to undergo treatment by either S-EMR or radiofrequency ablation(RFA). The initial staging EMR will not extend more than 50% of the esophageal circumference or more than 2 cm in longitudinal extent. Patients in the S-EMR group will undergo step-wise eradication of the BE segment using the Duette multi-band mucosectomy kit (Cook Medical, FDA approved) whereas those in the RFA group will undergo BE ablation using the endoscopically-guided HALO radiofrequency ablation system (Barrx Medical, FDA approved).

Both treatment groups will undergo their respective treatment sessions every 2 months until either no Barrett's esophagus is seen or until a maximum of 4 treatment sessions. Once there is no visible Barrett's esophagus, patients will undergo surveillance biopsies (random 4 quadrant biopsies every 1 cm of the neo-squamous mucosa and random biopsies of the cardia) to evaluate for complete eradication of Barrett's esophagus. Regardless of whether there is visible Barrett's esophagus, all patients will undergo repeat endoscopy every 2 months for 1 year after enrollment. If no visible Barrett's esophagus is seen during the endoscopy, then surveillance biopsies to evaluate for dysplasia will be taken. Regardless of whether this is any visible Barrett's esophagus, all patients will undergo surveillance biopsies at 12 months after enrollment.

The objective of this study is to compare the proportion of patients with complete eradication of Barrett's esophagus using S-EMR versus RFA at 12 months.

ELIGIBILITY:
Inclusion Criteria:

Subjects shall be screened according to the following inclusion criteria. An answer of "no" to any inclusion criterion disqualifies a subject from participating in this study.

* Patients age: > 18 years
* Subject has documented diagnosis of Barrett's esophagus, maximum endoscopic length of no more than C2M5 (i.e. no more than 2cm of circumferential extent and no more than 5cm of tongues) containing HGD/EC as follows:
* HGD or EC documented on biopsy within previous 6 months from enrollment
* Histology slides reviewed at central pathology service for ERADICATE Trial confirm HGD/EC.
* Endoscopically visible lesion/area/pattern in a patient with HGD/EC either by high definition white light endoscopy, narrow band imaging, confocal laser endomicroscopy, or another enhanced imaging tool.
* Ability to take oral proton pump inhibitor
* For female subjects of childbearing potential, a negative urine pregnancy test within 2 weeks of enrollment and any subsequent endoscopy encounter
* Subject is eligible for treatment and follow-up endoscopy and biopsy as required by the investigational plan
* Ability to discontinue aspirin/NSAIDs/Clopidogrel 7 days before and after all ablation procedures
* Ability of provide written, informed consent and understands the responsibilities of trial participation NOTE: At the Kansas City Veterans Hospital, participants must be eligible for care at the VA in order to be enrolled. Other sites listed are able to enroll non-veterans.

Exclusion Criteria:

Subjects shall be screened according to the following exclusion criteria. An answer of "yes" to any exclusion criterion disqualifies a subject from participating in this study.

* Extent of BE >C2M5
* The subject is pregnant or planning a pregnancy during the study period (12 months after treatment)
* Esophageal stricture preventing passage of endoscope or catheter
* Active erosive esophagitis
* History of malignancy of the esophagus, esophageal varices or coagulopathy
* Prior radiation therapy to the esophagus, except head and neck region radiation therapy.
* Any previous ablation therapy within the esophagus (photodynamic therapy, multipolar electrocoagulation, argon plasma coagulation, laser treatment, or other)
* Any previous EMR in the esophagus
* Any previous esophageal surgery, including fundoplication
* Evidence of esophageal varices during treatment endoscopy
* Subject has a life-expectancy of less than two years due to an underlying medical condition
* Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines
* Subject has an implantable pacing device (examples: Implantable cardiac defibrillator, neurostimulator, cardiac pacemaker) and has not received clearance for enrollment in this study by specialist responsible for the pacing device
* The subject is currently enrolled in an investigational drug or device trial that clinically interferes with the ERADICATE trial.
* Subject suffers from psychiatric or other illness deemed by the investigator as an inability to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Complete histological eradication of Barrett's esophagus | 12 months

SECONDARY OUTCOMES:
Complete histological clearance of dysplasia | 12 months
Complication rates | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Medical Center
Locations (3):
- United States (3):
  - University Of Chicago, Chicago, Illinois
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Columbia University, New York, New York

REFERENCES:
- [Background] Sharma P. Clinical practice. Barrett's esophagus. N Engl J Med. 2009 Dec 24;361(26):2548-56. doi: 10.1056/NEJMcp0902173. No abstract available. PMID 20032324
- [Background] Devesa SS, Blot WJ, Fraumeni JF Jr. Changing patterns in the incidence of esophageal and gastric carcinoma in the United States. Cancer. 1998 Nov 15;83(10):2049-53. PMID 9827707
- [Background] Sharma P, McQuaid K, Dent J, Fennerty MB, Sampliner R, Spechler S, Cameron A, Corley D, Falk G, Goldblum J, Hunter J, Jankowski J, Lundell L, Reid B, Shaheen NJ, Sonnenberg A, Wang K, Weinstein W; AGA Chicago Workshop. A critical review of the diagnosis and management of Barrett's esophagus: the AGA Chicago Workshop. Gastroenterology. 2004 Jul;127(1):310-30. doi: 10.1053/j.gastro.2004.04.010. PMID 15236196
- [Background] Buttar NS, Wang KK, Sebo TJ, Riehle DM, Krishnadath KK, Lutzke LS, Anderson MA, Petterson TM, Burgart LJ. Extent of high-grade dysplasia in Barrett's esophagus correlates with risk of adenocarcinoma. Gastroenterology. 2001 Jun;120(7):1630-9. doi: 10.1053/gast.2001.25111. PMID 11375945
- [Background] Reid BJ, Blount PL, Feng Z, Levine DS. Optimizing endoscopic biopsy detection of early cancers in Barrett's high-grade dysplasia. Am J Gastroenterol. 2000 Nov;95(11):3089-96. doi: 10.1111/j.1572-0241.2000.03182.x. PMID 11095322
- [Background] Weston AP, Sharma P, Topalovski M, Richards R, Cherian R, Dixon A. Long-term follow-up of Barrett's high-grade dysplasia. Am J Gastroenterol. 2000 Aug;95(8):1888-93. doi: 10.1111/j.1572-0241.2000.02234.x. PMID 10950031
- [Background] Heitmiller RF, Redmond M, Hamilton SR. Barrett's esophagus with high-grade dysplasia. An indication for prophylactic esophagectomy. Ann Surg. 1996 Jul;224(1):66-71. doi: 10.1097/00000658-199607000-00010. PMID 8678620
- [Background] Hulscher JB, van Sandick JW, de Boer AG, Wijnhoven BP, Tijssen JG, Fockens P, Stalmeier PF, ten Kate FJ, van Dekken H, Obertop H, Tilanus HW, van Lanschot JJ. Extended transthoracic resection compared with limited transhiatal resection for adenocarcinoma of the esophagus. N Engl J Med. 2002 Nov 21;347(21):1662-9. doi: 10.1056/NEJMoa022343. PMID 12444180
- [Background] Waxman I, Raju GS, Critchlow J, Antonioli DA, Spechler SJ. High-frequency probe ultrasonography has limited accuracy for detecting invasive adenocarcinoma in patients with Barrett's esophagus and high-grade dysplasia or intramucosal carcinoma: a case series. Am J Gastroenterol. 2006 Aug;101(8):1773-9. doi: 10.1111/j.1572-0241.2006.00617.x. Epub 2006 Jun 16. PMID 16780561
- [Background] Larghi A, Lightdale CJ, Memeo L, Bhagat G, Okpara N, Rotterdam H. EUS followed by EMR for staging of high-grade dysplasia and early cancer in Barrett's esophagus. Gastrointest Endosc. 2005 Jul;62(1):16-23. doi: 10.1016/s0016-5107(05)00319-6. PMID 15990814
- [Background] Inoue H, Endo M, Takeshita K, Kawano T, Goseki N, Takiguchi T, Yoshino K. Endoscopic resection of early-stage esophageal cancer. Surg Endosc. 1991;5(2):59-62. doi: 10.1007/BF00316837. PMID 1948615
- [Background] Giovannini M, Bories E, Pesenti C, Moutardier V, Monges G, Danisi C, Lelong B, Delpero JR. Circumferential endoscopic mucosal resection in Barrett's esophagus with high-grade intraepithelial neoplasia or mucosal cancer. Preliminary results in 21 patients. Endoscopy. 2004 Sep;36(9):782-7. doi: 10.1055/s-2004-825813. PMID 15326573
- [Background] Seewald S, Akaraviputh T, Seitz U, Brand B, Groth S, Mendoza G, He X, Thonke F, Stolte M, Schroeder S, Soehendra N. Circumferential EMR and complete removal of Barrett's epithelium: a new approach to management of Barrett's esophagus containing high-grade intraepithelial neoplasia and intramucosal carcinoma. Gastrointest Endosc. 2003 Jun;57(7):854-9. doi: 10.1016/s0016-5107(03)70020-0. PMID 12776032
- [Background] Peters FP, Kara MA, Rosmolen WD, ten Kate FJ, Krishnadath KK, van Lanschot JJ, Fockens P, Bergman JJ. Stepwise radical endoscopic resection is effective for complete removal of Barrett's esophagus with early neoplasia: a prospective study. Am J Gastroenterol. 2006 Jul;101(7):1449-57. doi: 10.1111/j.1572-0241.2006.00635.x. PMID 16863545
- [Background] Conio M, Repici A, Cestari R, Blanchi S, Lapertosa G, Missale G, Della Casa D, Villanacci V, Calandri PG, Filiberti R. Endoscopic mucosal resection for high-grade dysplasia and intramucosal carcinoma in Barrett's esophagus: an Italian experience. World J Gastroenterol. 2005 Nov 14;11(42):6650-5. doi: 10.3748/wjg.v11.i42.6650. PMID 16425359